CLINICAL TRIAL: NCT03753464
Title: The Role of Functional Epigenetic Modifications in Peri-Implantitis: A Pilot Clinical Study
Brief Title: The Role of Functional Epigenetic Modifications in Peri-Implantitis
Status: Completed | Type: Observational
Sponsor: NYU College of Dentistry (Other)
Responsible Party: Principal Investigator, Ismael Khouly, Clinical Assistant Professor, Department of Oral & Maxillofacial Surgery, NYU College of Dentistry
Other Study IDs: 18-00986
Record Dates: First submitted 2018-11-15; First posted 2018-11-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Periimplantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gingival and blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peri-implantitis: Patients undergoing surgical treatment for peri-implantitis. Gingival and blood samples will be collected during the treatment for peri-implantitis.
  Interventions: Procedure: Gingival biopsy and blood sample collection
- Healthy: Healthy patients undergoing treatment for either wisdom tooth extraction or gingivectomy. Gingival and blood samples will be collected during either wisdom tooth extraction or gingivectomy.
  Interventions: Procedure: Gingival biopsy and blood sample collection

INTERVENTIONS:
Procedure: Gingival biopsy and blood sample collection — Gingival and blood samples will be collected.

SUMMARY:
The aim of this pilot, exploratory, single blind clinical trial is to evaluate the epigenetic changes associated with peri-implantitis.

DETAILED DESCRIPTION:
Twenty patients will be voluntarily enrolled in two groups: 10 healthy participants, and 10 participants with peri-implantitis. Periodontal and peri-implant clinical and radiographic measurements, as well as body mass index, medical and dental history will be recorded within the following timelines: at baseline (for both groups), and 6 months after baseline for the peri-implantitis group only. At baseline, gingival biopsies and blood will be harvested from: a) healthy gingival sites during either surgical removal of wisdom teeth or gingivoplasty, in the healthy group; and, b) from a peri-implantitis site during surgical treatment of peri-implantitis, and when possible, from a healthy gingival site within the same participant, in the peri-implantitis group. After harvesting of biopsies, peri-implantitis subjects will be re-evaluated 6 months after treatment. During the 6-month visit, if a second surgical treatment of peri-implantitis in the same implant treated at baseline is indicated as standard of care of the participant, a new gingiva biopsy and blood will be collected. Gingival biopsies and blood collected from each participant will be used to perform DNA methylation analysis.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Subjects must have read, understood, and signed an informed consent form.
* Subjects must be 20-90 years of age.
* Subjects must be non-smokers or ex-smokers who have quit smoking for at least one year prior to enrollment in the study.
* Subjects must be in good general health as assessed by the Investigator.

Healthy Periodontal Subjects Inclusion Criteria:

In addition to the general inclusion criteria, a healthy periodontal subject must meet all of the following criteria:

• Subjects show gingival health and no history of periodontitis, as described in the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions.

Peri-implantitis Subjects Inclusion Criteria:

In addition to the general inclusion criteria, a PIT subject must meet all of the following criteria:

* Subjects with implant-supported prosthesis/es in function for at least 12 months who had at least one implant diagnosed with peri-implantitis based on the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions.
* Subjects must be committed to the study and the required follow-up visits.
* Standard of care treatment of the diseased implant with PID will consist on open flap debridement (OFD).

Exclusion Criteria:

General Exclusion Criteria:

* Pregnant or lactating.
* Use of antibiotics, within 1 month before enrollment in the study.
* Chronic use of nonsteroidal anti-inflammatory drugs for over 3 weeks of continuous use at the time of enrollment or during the course of the study.
* Requirement for prophylactic antibiotics for dental procedures.
* Mucosal diseases in the localized area around the biopsy site.
* Subjects with a systemic disease that would preclude biopsy/oral surgery.
* History of local irradiation therapy in the head/neck area.
* Subjects with poor oral hygiene.
* Subjects receiving, or having a history of receiving intravenous or subcutaneous anti-resorptive agents associated with osteonecrosis of the jaw.
* Subjects with any untreated endodontic lesions or untreated periodontal disease adjacent to the biopsy site.
* Acute necrotizing ulcerative gingivitis or gross tooth decay, as determined by the investigator.
* Subjects with conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis.

Periodontally Healthy Subjects Exclusion:

In addition to the general exclusion criteria, subjects allocated to the healthy group who meet any of the following criteria will be excluded from participation in this study:

• Root fragments, pericoronitis, endo-perio lesions, gross tooth decay, or other dental abscesses at the biopsy site. Subjects may be rescreened after resolution of these dental conditions.

Peri-implantitis subjects Exclusion:

In addition to the general exclusion criteria, subjects allocated to the PIT group who meet any of the following criteria will be excluded from participation in this study:

* Inadequate implant position (i.e., prosthetically driven).
* PIT due to excess of cement.
* Subjects who have physical or mental handicaps that would interfere with the ability to perform adequate oral hygiene.
* Subjects with implants previously surgically treated for PIT.
* Less than 2mm of keratinized peri-implant tissue.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Periodontally Healthy Subjects
  * Peri-implantitis Subjects
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Differences in epigenetic signatures in peri-implantitis subjects as compared to healthy subjects, in an exploratory manner. (Gingival biopsies and blood collected to perform DNA methylation analysis) | 6 months
  Gingival and blood samples collected from healthy subjects and subjects with peri-implantitis will be used to determinate epigenetic signatures associated with peri-implantitis.
Epigenetic signatures associated with response to treatment peri-implantitis at 6 months, in an exploratory manner. (Differences in epigenetic signatures in peri-implantitis subjects as compared to healthy subjects, in an exploratory manner. | 6 months
  Samples collected from patients with peri-implantitis will be used to determinate epigenetic signatures associated response to treatment peri-implantitis at 6 months. (Gingival biopsies and blood collected to perform DNA methylation analysis)

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) will be assessed to determinate patient-reported outcome measures, at baseline and at 6 months. | 6 months
  A visual analog scale (VAS) will be used to evaluate patient's pain/discomfort, esthetic satisfaction, and the subjects' overall satisfaction at baseline and at 6 months.
Oral Health Impact Profile-14 (OHIP-14) will be assessed to determinate patient-reported outcome measures, at baseline and at 6 months. | 6 months
  Oral Health Impact Profile-14 (OHIP-14) assessed at baseline and at 6 months.
Changes in peri-implant pocket depths (PPD) (in mm) from baseline to 6 month after surgery (only peri-implantitis group). | 6 months
  Peri-implant pocket depths (PPD) will be assessed at baseline and 6 month after surgery.
Changes in peri-implant BOP (in percentage), from baseline to 6 month after surgery (only peri-implantitis group). | 6 months
  Peri-implant BOP (in percentage) will be assessed at baseline and 6 month after surgery.
Percentage of peri-implant pocket closure at to 6 month after surgery (only peri-implantitis group). | 6 months
  Percentage of peri-implant pocket closure will be assessed at at to 6 month after surgery.
Changes in peri-implant marginal bone level (in mm) from baseline to 6 month after surgery (only peri-implantitis group). | 6 months
  Mean crestal bone level change around the implants will be determined by periapical radiographs of mesial and distal bone levels from baseline to 6 months surgery.
Change in soft tissue levels (in mm) from baseline to 6 month after surgery (only peri-implantitis group). | 6 months
  Soft tissue levels assessed at baseline and 6 months post-surgery in implants with peri-implantitis.
Incidence of post-operative surgical site infections (only peri-implantitis group). | 6 months
  Number of post-operative surgical site infections from surgery to 6 months.
Incidence of post-operative complications (only peri-implantitis group). | 6 months
  Number of post-operative complications from surgery to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Khouly, DDS, MS, PhD, Principal Investigator — New York University
Locations (1):
- Bluestone Center for Clinical Research. New York University College of Dentistry, New York, New York, United States